CLINICAL TRIAL: NCT01626677
Title: Long Term Follow-Up Study of CARTISTEM® Versus Microfracture for the Treatment of Knee
Brief Title: Follow-Up Study of CARTISTEM® Versus Microfracture for the Treatment of Knee Articular Cartilage Injury or Defect
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARTISTEM_CR_F/U; NCT01923532 (obsolete NCT alias)
Record Dates: First submitted 2012-06-19; First posted 2012-06-25 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Degenerative Osteoarthritis; Defect of Articular Cartilage
Keywords: Umbilical Cord Blood; Mesenchymal Stem Cells; Cartilage injury; Osteoarthritis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARTISTEM (Experimental): A single dose of 500㎕/㎠ of cartilage defect
  Interventions: Biological: CARTISTEM
- Microfracture (Active Comparator): conventional treatment method
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Biological: CARTISTEM — A single dose of 500㎕/㎠ of cartilage defect
  Other Names: hUCB-MSCs
  Arms: CARTISTEM
Procedure: Microfracture — Active control
  Other Names: Conventional surgical treatment
  Arms: Microfracture

SUMMARY:
This is a long term follow-up study to investigate the safety and efficacy of CARTISTEM®, human umbilical cord blood-derived mesenchymal stem cells, in repair of cartilage injury or defects, compared with microfracture. Subjects who participated in and completed the Phase III trial (NCT01041001) will be tracked until the 60 month post-treatment timepoint.

DETAILED DESCRIPTION:
This long term follow-up study is performed to assess the long-term safety and efficacy of CARTISTEM®, human umbilical cord blood-derived mesenchymal stem cells, in repair of cartilage injury or defects, compared with microfracture. Subjects, who were either administered CARTISTEM or treated with conventional microfracture in the primary phase III study (NCT01041001), will be further observed using various subjective knee assessments and MRI T2 mapping until the 60 month post-treatment timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee joint cartilage defect or injury of ICRS (International Cartilage Repair Society) Grade 4 confirmed by arthroscopy (At screening, patients diagnosed as such with an MRI may be included)
* Male or female patients at least 18 years of age
* Patients whose lesion (unilateral joint) is 2 ㎠ ~ 9㎠ in size
* Patients with articular swelling, tenderness and active range of motion of Grade 2 or below
* Patients with pain in affected joint of 60-mm or below on a 100-mm VAS (visual analogue scale)
* Patients with adequate blood coagulation activity: PT(INR) < 1.5, APTT <1.5×control
* Patients with adequate renal function: Creatinine ≤ 2.0 ㎎/㎗, levels of proteinuria measured with Dipstick: trace or less
* Patients with adequate hepatic function: Bilirubin ≤ 2.0 ㎎/㎗, AST/ALT ≤ 100 IU/L
* Patients who have received no surgery or radiation therapy in the affected joint within the past 6 six weeks, and have recovered from the side effects of such past treatments
* Female patients of childbearing potential must agree to practice adequate methods of birth control to prevent pregnancy during the study
* Patients whose physical examination results show no ligament instability of Grade II or above (Grade 0: none, Grade I: 0-5 mm, Grade II: 5-10 mm, Grade III: >10 mm)
* Patients who voluntarily agreed to enroll in the study and signed an informed consent form

Exclusion Criteria:

* Patients with autoimmune disease or the medical history
* Patients with infections requiring parenteral administration of antibiotics
* Patients with myocardial infarction, ischemic heart failure, other serious heart conditions or uncontrolled hypertension, or any medical history of such diseases
* Patients with serious internal diseases
* Patients who are currently pregnant or nursing
* Patients with psychotic diseases, epilepsy, or any history of such diseases
* Patients with alcohol abuse
* Patients who smoke excessively
* Patients with chronic inflammatory articular diseases such as rheumatoid arthritis
* Patients who were enrolled in any other clinical trials within the past four weeks
* Patients who had been administered with immunosuppressants such as Cyclosporin A or azathioprine within the past six weeks
* Patients whose physical examination results show ligament instability of Grade II or above (Grade 0: none, Grade I: 0-5 mm, Grade II: 5-10 mm, Grade III: >10 mm)
* Patients with a known history of hypersensitivity/allergy to gentamicin
* Patients whom the principal investigator considers inappropriate for the clinical trial due to any other reasons than those listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Degree of improvement in knee assessments compared to the active control (microfracture) | 36 months, 48 months, and 60 months
  Knee assessments will be performed using the following tools:
  * IKDC (International Knee Documentation Committee)
  * Pain score on VAS (Visual Analogue Scale)
  * WOMAC (Western Ontario and McMaster Universities Arthritis Index)

SECONDARY OUTCOMES:
Number of subjects with adverse events | 36 months, 48 months, and 60 months
  Systemic and local adverse events especially attributable to the implanted cells will be assessed.
  * General physical examinations: vital signs, blood tests
  * Physical assessments of the knee: swelling, tenderness, pain, range of motion
  * Tumor formation at the implantation site: radiological evaluation using MRI(T1(dGEMRIC)and T2 mapping)

CONTACTS AND LOCATIONS:
Overall Officials: Hong-chul Lim, MD, PhD, Principal Investigator — Korea University Guro Hospital; Beom-gu Lee, MD, PhD, Principal Investigator — Gachon University Gil Medical Center; Jong-hyeok Choi, MD, PhD, Principal Investigator — Gangnam Severance Hospital; Hwa-jae Jeong, MD, PhD, Principal Investigator — Kangbuk Samsung Hospital; Chul-won Ha, MD, PhD, Principal Investigator — Samsung Medical Center; Jung-ro Yoon, MD, PhD, Principal Investigator — Seoul Veterans Hospital; Seong-il Bin, MD, PhD, Principal Investigator — Asan Medical Center; Jae-doo Yoo, MD, PhD, Principal Investigator — Ewha Womans Mokdong Hospital; Myung-ku Kim, MD, PhD, Principal Investigator — Inha University Hospital; Choong-hyuk Choi, MD, PhD, Principal Investigator — Hanyang University; Young-Chul Yoon, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (10):
- South Korea (10):
  - Inha University Hospital, Incheon
  - Gachon University Gil Hospital, Incheon
  - Kangbuk Samsung Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Seoul Veterans Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lim HC, Park YB, Ha CW, Cole BJ, Lee BK, Jeong HJ, Kim MK, Bin SI, Choi CH, Choi CH, Yoo JD; Cartistem Research Group; Yoon JR, Chung JY. Allogeneic Umbilical Cord Blood-Derived Mesenchymal Stem Cell Implantation Versus Microfracture for Large, Full-Thickness Cartilage Defects in Older Patients: A Multicenter Randomized Clinical Trial and Extended 5-Year Clinical Follow-up. Orthop J Sports Med. 2021 Jan 12;9(1):2325967120973052. doi: 10.1177/2325967120973052. eCollection 2021 Jan. PMID 33490296
- See also: Study to Compare the Efficacy and Safety of Cartistem® and Microfracture in Patients With Knee Articular Cartilage Injury or Defect — http://clinicaltrials.gov/ct2/show/NCT01041001?term=cartistem&rank=1